CLINICAL TRIAL: NCT00778648
Title: Effectiveness of an Encapsulated Juice Powder Concentrate for Preventing Common Cold Symptoms
Brief Title: Encapsulated Juice Powder Concentrate for Preventing Common Cold Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NSA, Collierville, TN, USA (Unknown)
Responsible Party: Institute for Social Medicine, Epidemiology & Health Economics, Charite University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JPCC
Record Dates: First submitted 2008-10-21; First posted 2008-10-23 (Estimated); Results first posted 2010-10-05 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-09

CONDITIONS: Common Cold
Keywords: Common cold; prevention; dietary supplement
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Juice Plus (Experimental)
  Interventions: Dietary Supplement: Juice Plus
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Juice Plus — Juice Plus+® is a dietary supplement from concentrated fruits (apple, orange, pineapple,cranberry, cherry (acerola), papaya and peach) and vegetables (carrot, parsley, beet, broccoli, kale, cabbage, spinach, and tomato).
  Subjects will take four capsules of Juice Plus+® daily.
  Other Names: Juice Plus+®
  Arms: Juice Plus
Dietary Supplement: Placebo — Four capsules of placebo daily.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the effect of an encapsulated juice powder concentrate on the number of days with at least moderate common cold symptoms over winter time.

DETAILED DESCRIPTION:
Common cold is the most frequent acute illness in industrialised societies. Though it is usually benign, it is a leading cause of absence from work and doctor visits, causing an enormous economic burden including lost productivity and treatment costs.

Common cold is caused by a variety of viruses, with rhinoviruses and corona viruses as the most common. There is currently no treatment for common cold, thus therapy is focussed on symptom relief only. Prevention strategies for common cold include lifestyle measures such as avoiding infected people and regular hand washing during cold season. Dietary supplements including herbs and vitamins have been suggested as preventive strategies for common cold.

Juice Plus+® is a dietary supplement composed primarily of juice powder concentrate and pulp from fruits and vegetables. It contains several antioxidants including vitamin C, vitamin E, beta-carotene and folate. One randomized study reported reduction in work days lost to illness in the Juice Plus+® group compared to the placebo group. However, the clinical benefit for preventing common cold symptoms has not yet been tested in a large adult population.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 18-65 years of age.
* Able and willing to take the active or placebo capsules over the whole study period.
* Health care professionals with essential patient contact (physicians, nurses, physiotherapists, etc) in Berlin, Germany.
* Written informed consent.

Exclusion Criteria:

* Known or suspected hypersensitivity or allergy to one of the ingredients of Juice Plus+®.
* Refusal to stop intake of additional vitamin supplements during study.
* Pregnancy or Lactation.
* Alcohol addiction, drug abuse or any other condition considered by the investigator to interfere with study procedures.
* Language limitations regarding interviews and questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan N. Willich, Prof, Principal Investigator — Institute for Social Medicine, Epidemiology & Health Economics
Locations (1):
- Institute for Social medicine, Epidemiology & Health Economics, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Lamprecht M, Oettl K, Schwaberger G, Hofmann P, Greilberger JF. Several indicators of oxidative stress, immunity, and illness improved in trained men consuming an encapsulated juice powder concentrate for 28 weeks. J Nutr. 2007 Dec;137(12):2737-41. doi: 10.1093/jn/137.12.2737. PMID 18029492

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Juice Plus | Placebo
Started | 272 | 271
Completed | 263 | 266
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Juice Plus | Placebo | Total
Number analyzed (Participants) | 272 | 271 | 543
Age Continuous [Mean (Standard Deviation); unit: years] | 40.9 (10.2) | 38.8 (10.3) | 40.9 (10.2)
Gender [Number; unit: participants]
  Female | 202 | 222 | 424
  Male | 61 | 44 | 105
Region of Enrollment [Number; unit: participants]
  Germany | 272 | 271 | 543

OUTCOME MEASURES:

1. Primary Outcome: Number of Days With at Least Moderate (i.e. Moderate or Severe) Common Cold Symptoms.
Time Frame: within 6 months (after 2 months run-in period)
Measure: Mean (95% Confidence Interval); unit: Number of days
Arm/Group | Juice Plus | Placebo
Number analyzed (Participants) | 272 | 271
Number of days | 7.6 [6.5 to 8.8] | 9.5 [8.4 to 10.6]
Statistical Analysis 1: Comparison: Juice Plus vs Placebo; Test type: Superiority or Other; p = 0.023, ANOVA

2. Secondary Outcome: Secondary Endpoints of This Study Are Mean Health-related Quality of Life, Mean Common Cold Related Total Costs, Direct and Indirect (Productivity Loss) Costs
Time Frame: Baseline, months 2,4,6,8.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Juice Plus | Placebo
Serious Adverse Events (participants affected / at risk) | 0/272 | 0/271
Other Adverse Events (participants affected / at risk) | 0/272 | 0/271

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No